CLINICAL TRIAL: NCT04785066
Title: Evaluation of the Efficacy of Dornase Alfa (Pulmozyme®) on Arterial Recanalization in Post-thrombectomy Angiography in Patients With Ischemic Stroke by Thrombolysis and Eligible for Thrombectomy (NETs-target)
Brief Title: Efficacy of Pulmozyme® on Arterial Recanalization in Post-thrombectomy Patients Managed for Ischemic Stroke (NETs-target)
Acronym: NETs-target
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDS_2021_5
Record Dates: First submitted 2021-02-23; First posted 2021-03-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Administration of dornase alfa during intervention of thrombectomy
  Interventions: Drug: Administration of dornase alfa

INTERVENTIONS:
Drug: Administration of dornase alfa — Patient treated for a cerebral thrombectomy will be administred dornase alfa treatment by intravenous

SUMMARY:
The functional prognosis of patients with ischaemic stroke treated by thrombolysis and thrombectomy is associated with complete reperfusion of the occluded artery defined by an mTICI 2C or 3 score at the end of thrombectomy. However, this complete reperfusion is only obtained in 60% of patients. Most often, incomplete reperfusion is due to the persistence of distal occlusions, which are inaccessible to mechanical thrombectomy. Drug treatment, combined with thrombectomy to increase the rate of complete reperfusion, would be a major advance in the management of these patients.

This is a non-randomized, monocentric, open-label, phase II trial to evaluate efficacy of dornase alfa intravenous administration in patients treated with intravenous thrombolysis and eligible for thrombectomy for ischemic stroke of the anterior circulation.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke by proximal intracranial occlusion (internal carotid artery, middle cerebral artery in its M1 or M2 segment) isolated from the anterior circulation eligible for cerebral thrombectomy.
* Transferred to the NRI block for a cerebral thrombectomy.
* Treated by thrombolysis intravenous (Aleplase or Tenecteplase) as recommanded by European stroke organisation
* With DWI-ASPECT score>5 to MRI

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Known allergy to Dornase alfa or one of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of intravenous administration of dornase alfa (Pulmozyme®) on arterial recanalization in post-thrombectomy patients managed for ischemic stroke | 3 months after procedure
  Complete recanalization defined by a modified treatment in cerebral infarction (mTICI) 2C or 3 score at cerebral angiography one hour after the start of pulmozyme administration or at the end of the thrombectomy procedure (if procedure >1h).
  * The grade 2C corresponds to : Near complete perfusion except for slow flow in a few distal cortical vessels, or presence of small distal cortical emboli.
  * The grade 3 corresponds to: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Paris, France